CLINICAL TRIAL: NCT02803359
Title: Investigation of Human Laryngeal Evoked Brainstem Potentials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-414
Record Dates: First submitted 2016-06-06; First posted 2016-06-17 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Thyroidectomy
Keywords: Laryngeal evoked brainstem response (LEBR); laryngopharyngeal sensory discrimination testing (LPSDT); brainstem activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Planned Procedure (Experimental): Endoscope will be connected to a camera and monitor. Needle electrodes will then be positioned into the false vocal fold mucosa bilaterally, under direct visualization of the needle tip on the monitor, but the needles will be passed trans-orally in the operating room. For those participating during an open-neck surgery, the surgery will commence as planned and once exposure of the superior laryngeal nerve is obtained, the surgeon will insert the electrodes directly into the nerve trunk for the purposes of recording. In Surgery or cervical lymphadenectomy, the electrode will be placed at a superficial depth and needle placement will be performed with one on each side at a location approximately mid-fold.
  Interventions: Procedure: Placement of a needle electrode through the thyrohyoid membrane into the submucosal space within the false vocal fold
- Routine Laryngoscopy (Experimental): Nasolaryngoscopy will be performed in the office in the standard fashion with the use of oxymetazoline for topical decongestion of the nasal mucosa, In both settings, the electrode will be placed at a superficial depth and needle placement will be performed with one on each side at a location approximately mid-fold
  Interventions: Procedure: Placement of a needle electrode through the thyrohyoid membrane into the submucosal space within the false vocal fold

INTERVENTIONS:
Procedure: Placement of a needle electrode through the thyrohyoid membrane into the submucosal space within the false vocal fold

SUMMARY:
The primary purpose of this study will be to determine whether the proposed study protocol will allow for reliable detection of the human Laryngeal evoked brainstem responses (LEBR). Laryngeal evoked brain stem responses will be recorded from five test subjects under general anesthesia in the operating room with the assistance of an electrophysiologist with expertise in evoked potentials. Once the feasibility of obtaining tracings are established on the first few subjects, responses will be recorded from other test subjects with the aim of determining the optimal placement of stimulating electrodes and detection leads necessary to elicit an adequate response. The effect of varying the stimulus intensity will also be studied. Once parameters for testing have been standardized, normative configurations for the laryngeal evoked brainstem response tracings can be determined by patients both in the office setting and in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects undergoing thyroid or other open neck surgeries

Exclusion Criteria:

* Current or recent (within one month) tracheostomy
* Vocal cord paralysis
* History of Stroke
* History of Diabetes Mellitus
* History of Neurologic Disease
* History of Radiation to the Neck
* History of Brain Surgery
* History of Neck Surgery
* Recent Laryngeal Surgery (within one month)
* Recent Intubation (within two weeks)
* Laryngopharyngeal Reflux Disease
* Allergy to Lidocaine
* Allergy to Oxymetazoline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-06; Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
analysis of variance in brain auditory evoked response (BAER) measured using recording electroencephalography electrodes | One Year
  Distributions of latencies within this group will be examined to evaluate the appropriateness of standard assumptions regarding normality and constant variance, and transformations or non-parametric statistics will be considered as needed.

CONTACTS AND LOCATIONS:
Overall Officials: Milan Amin, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States